CLINICAL TRIAL: NCT00825760
Title: Phase II Randomised, Placebo Controlled Trial to Investigate Repeat Dose Antimicrobial Photodynamic Therapy in Patients With Chronic Leg Ulcers.
Brief Title: Clinical Trial to Investigate Treatment With Photodynamic Therapy to Reduce Levels of Bacteria in Leg Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Photopharmica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PPA/904W/003
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Chronic Leg Ulcers; Wound Healing
Keywords: Antimicrobial Photodynamic Therapy; Photodynamic Therapy; PDT; Red light; Visible light; Antimicrobial; Antibacterial; Wound healing; Wound management; Leg ulcer; Chronic venous leg ulcer; Chronic wound; Wound therapy; Antimicrobial therapy
MeSH Terms: conditions — Leg Ulcer | interventions — Light

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): Single treatment
  Interventions: Drug: Topical PPA904 gel and light; Drug: Topical placebo gel plus light
- 2 (Other): 12 treatments, once weekly
  Interventions: Drug: Topical PPA904 gel and light; Drug: Topical placebo gel plus light

INTERVENTIONS:
Drug: Topical PPA904 gel and light
Drug: Topical placebo gel plus light

SUMMARY:
Some leg ulcers do not seem to respond that well to the standard treatments that we currently use. One reason for this may be that there are high levels of bacteria in the ulcer which may be slowing down the rate of healing. Because we need to be careful about when we use antibiotics, this study will look at another way of killing bacteria in the ulcer. This new method involves putting a special gel on the ulcer and then shining a particular type of light (visible red light) onto the ulcer for a short period of time.

In the first part of the study, a single treatment with the gel and light will be investigated. The second part of the study will compare whether or not using the treatment once a week for 12 weeks is better than placebo.

Across the UK 57 people with chronic leg ulcers will be asked to take part in this study (9 in part 1 and 48 in part 2). Up to 10 sites will be involved including Cardiff University and hospitals in Bradford, Harrogate, Dundee, Hull, Plymouth and the Wirral.

The research is funded by Photopharmica Ltd.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be males or females of non-childbearing status over 18 years of age.
* Subjects will have a chronic leg ulcer with an ABPI ≥ 0.6 (measured at screening).
* Subjects will have an ulcer that has been present for at least 3 months and not more than 3 years.
* Subjects will have an ulcer with an area of 2 - 100cm2 and a maximum linear dimension of 10cm.
* Subjects will have an ulcer with a total bacterial load of ≥ 104 CFU / cm2, determined within 2 weeks before the first treatment.
* Subjects will have voluntarily signed and dated a subject Informed Consent Form (ICF).
* Subjects will be, in the opinion of the Investigator, able to understand the study, co-operate with the study procedures and be willing to return to the clinic for all the required follow-up visits.
* Subjects should be of appropriate health to participate in the study, as determined by the Investigator. This will be determined by a medical history, physical examination, 12-lead ECG and clinical laboratory evaluations.

Exclusion Criteria:

* Subjects under the age of 18 years of age.
* Subjects who have taken topical or systemic antibiotics during the 2 weeks prior to screening.
* Subjects who have used any anti-microbial dressing or topical antiseptic / antimicrobial or received maggot therapy during the 2 weeks prior to screening.
* Subjects who have evidence of connective tissue disorders e.g. vasculitis or rheumatoid arthritis under active treatment.
* Subjects who have any clinically significant medical condition that would impair wound healing as determined by the investigator, including uncontrolled diabetes as determined by HbA1C (>12%) or immune disease.
* Subjects who are known to abuse alcohol or drugs currently, or to have psychological disorders that could affect follow-up care or treatment outcomes.
* Subjects who have received short course corticosteroids within 30 days prior to treatment.
* Subjects who have participated in a clinical trial of any investigational drug within 4 months prior to treatment.
* Subjects who have participated in a clinical trial of any investigational device, for example dressings, within 1 month prior to treatment.
* Subjects who have previously been treated with IMP in this trial.
* Subjects who have or are suspected of having malignancy, or who have received treatment for any active malignancy, apart from non-melanomatic skin cancer, within 3 months prior to treatment.
* Subjects with evidence of exposed bone, tendon or facia visible around the target wound.
* Subjects with photosensitivity disorders.
* Subjects with systemic infection, whether or not related to their ulcer.
* Subjects with clinically relevant (assessed by PI) active wound infection undergoing treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2009-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To determine if repeat dose antimicrobial photodynamic therapy with PPA904 and PPA Lux 680 can cause a reduction in the bacterial content of chronic leg ulcers. | Measurement of total bacterial load of the ulcer immediately before and after each treatment.

SECONDARY OUTCOMES:
Measurement of the levels of specific bacteria, including anaerobes, S.aureus (MSSA and MRSA), P.aeruginosa and beta-haemolytic Streptococci in the ulcer. | Immediately before and after each treatment.
Measurement of the ulcer area. | Weekly for 12 weeks post the first dose compared to pre the first dose for subjects receiving 12 doses (part 2 of the study).
Assessment of pain. | Pre the first dose and weekly for 12 weeks post the first dose for subjects receiving 12 doses (part 2 of the study).
Assessment of quality of life using the Cardiff Wound Impact Schedule | Pre the first dose and 12 weeks post the first dose for subjects receiving 12 doses (part 2 of the study).
Measurement of PPA904 levels in peripheral blood samples. | Pre-dose and 1h, 3h and 24h post-dose for subjects receiving 1 dose (part 1 of the study).
Safety parameters including: vital signs, 12 lead ECG, blood and urine samples, physical examination and adverse event questioning. | 24 hours for subjects receiving 1 dose (part 1 of the study). 6 and 12 weeks post first dose for subjects receiving 12 doses (part 2 of the study).

CONTACTS AND LOCATIONS:
Overall Officials: Keith Harding, MBChB FRCS, Principal Investigator — Cardiff University
Locations (4):
- United Kingdom (4):
  - Department of Vascular Surgery, Bradford Royal Infirmary, Bradford
  - Department of Wound Healing, Cardiff University, Cardiff
  - Dermatology Department, Ninewells Hospital and Medical School, Dundee
  - Dermatology Department, Harrogate District Hospital, Harrogate

REFERENCES:
- See also: The 'Wound Healing Research Unit, Cardiff University' is a collaborator for this study, — http://www.whru.co.uk/